CLINICAL TRIAL: NCT01992666
Title: GENetic & Immunologic Abnomalies in Systemic Lupus Erythematosus
Acronym: GENIAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012.769; 2012-A01449-34 (Other: ID-RCB)
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic lupus erythematosus; genetic; immunological; pediatric; mutation; lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood sampling (Experimental)
  Interventions: Genetic: Blood sampling

INTERVENTIONS:
Genetic: Blood sampling — Immunologic and genetic analysis from a single blood sample.

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease for which the aetiology includes genet-ic and environmental factors. It is rare in children as compared to adults. The severity may be related to greater involvement of genetic factors in children. The impact of genetics in the development of SLE is important, and the risk of recurrence in siblings evaluated by lambda S ratio is 30 in SLE, while it is 15 for type-1 diabetes and 8 rheumatoid arthritis, thereby indicating high impact of genetics in SLE.

Recently, the group of Professor Yanick Crow in Manchester and other teams has identified new forms of lupus Mendelian genetics. The TREX1 and genes involved in the SAMHD1 frostbite lupus.

Nearly 2 % of all adult subjects with SLE have a heterozygous mutation in the TREX1 gene, which therefore represents the first genetic cause of SLE. The team of Professor Crow also identified the ACP5 gene that is responsible for SLE associated with Spondylo-epiphyseal enchondro-epiphyseal dysplasia (syndromic lupus). Other groups have identified mutations in two genes encoding a DNAse (DNAse1 and DNAse1L3) responsible for familial monogenic forms of SLE. These new genes SLE were identified through research of germ-line mutations in cases of lupus syndromic or family. In collaboration with Professor Crow, we are currently undergoing characterization of a novel gene of SLE in a family and we have identified a second locus identified in another family. The identification of these genes provides a better understanding of the mechanisms regulating immune tolerance in humans. The frequency of these genetic forms is not known. There is very little data on the immunological phenotype of these patients.

This is a clinical study to investigate the genetic and immunological abnormalities associated with pediatric SLE. The aim are to:

* study the genetics of pediatric SLE (or syndromic or family) and to search for mutations in the known genetic lupus or new genes in collaboration with Professor Yanick Crow.
* study the lymphocyte subpopulations and serum cytokines in pediatric patients with SLE (or syndromic or family) in the large Rhône- Alpes- Auvergne area.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, major or minor of any age with SLE (defined according to the ACR criteria)

   * Onset pediatric (<18 years) OR
   * Syndromic Lupus (associated with growth retardation, neurological deficit not related to lupus, frostbite, lymphoproliferation, the kidney malformations, heart, lung, brain calcifications) OR
   * Lupus in context with familial consanguinity OR
   * Familial cases (2 cases of SLE related first degree relative) OR related topic of the first degree to a lupus patient participant (if family lupus or related parents) OR
   * mother/father's lupus patient (in cas of simplex lupus)
2. A person or beneficiary entitled to a social security scheme or similar
3. Informed consent signed by the person (or parent / holding parental authority for minors)

Exclusion Criteria:

- none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
New genes identification | Once. At inclusion.
  Description: Identification of genetic mutations in the following genes: TREX1, SAMHD1, ACP5, DNAse1, DNAse1L3, or in new lupus genes.

SECONDARY OUTCOMES:
Immunological genotype and clinical abnormalities correlation | Once. At inclusion
  Correlate genotype to immunological (interferon alpha, …) and clinical abnormalities (microcrania, growth retardation, …)

OTHER OUTCOMES:
Immunological component | Once. At inclusion
  Identification of specific immunological factors of pediatric patients with SLE (or syndromic or family)
Characterization of sub-groups: size, articular manifestations (SLEDAI), hematology (hemoglobin, platelets, G White, ANA, ds-DNA, C3, C4, CH50, creatinine, proteinuria. | Once. At inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Belot, Dr, Study Director — Hospices Civils de Lyon
Locations (26):
- France (26):
  - Service d'hématologie / oncologie pédiatrique - CHU, Angers
  - Néphrologie Pédiatrique - CHU Besançon, Besançon
  - Hôpital Femme Mère Enfant, Bron
  - Service de Néphrologie Pédiatrique, Clermont-Ferrand
  - Service de pédiatrie - CHU Fort de France, Fort de France
  - Service de Néphrologie et Rhumatologie Pédiatrique, Grenoble
  - Service de Rhumatologie Pédiatrique - Hôpital de Bicêtre, Le Kremlin-Bicêtre
  - Service de médecine interne - Centre de référence des maladies rares, Lille
  - Service de néphrologie, endocrinologie, maladie métabolique et hématologie bénigne pédiatriques - Hôpital Jeanne de Flandre, Lille
  - édiatrie générale, urgences et maladies infectieuses, Hôpital Salengro, Lille
  - Service de Néphrologie - Hôpital Edouard Herriot, Lyon
  - Centre de néphrologie et de transplantation rénale - Hôpital de la conception, Marseille
  - Service de médecine infantile- Hôpital Nord, Marseille
  - Service de médecine interne - Hôpitaux privés de Metz, Metz
  - ervice d'urgence et post-urgences pédiatriques - CHU Arnaud de Villeneuve, Montpellier
  - Service médecine infantile 2, Nancy
  - Service de néphrologie pédiatrique - CHU de Nantes, Nantes
  - Service d'immunologie et rhumatologie pédiatrique - Centre de référence de maladies rhumatologiques et inflammatoires rares en pédiatrie-Hôpital Necker-Enfants malades, Paris
  - Service de médecine interne - Hôpital Saint Antoine, Paris
  - Service de pédiatrie générale - Hôpital Robert-Debré, Paris
  - Médecine Interne Adulte - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service de Rhumatologie - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Service pédiatrie grands enfants-adolescents - CHU Hôpital Sud, Rennes
  - Hôpital Nord, Saint-Etienne
  - Service de Pédiatrie Générale - CHU Réunion, Saint-Pierre
  - Service de néphrologie - médecine interne - Hypertension pédiatrique - Hôpital des enfants, Toulouse

REFERENCES:
- [Result] Weill O, Decramer S, Malcus C, Kassai B, Rouvet I, Ginhoux T, Crow YJ, Rieux-Laucat F, Soulas-Sprauel P, Pagnier A, Kone-Paut I, Piram M, Galeotti C, Samaille C, Reumaux H, Lanteri A, Dubois SM, Lefebvre H, Burtey S, Maurier F, Carbasse A, Lemelle I, Meinzer U, Despert V, Flodrops H, Fabien N, Ranchin B, Hachulla E, Bader-Meunier B, Belot A. Familial and syndromic lupus share the same phenotype as other early-onset forms of lupus. Joint Bone Spine. 2017 Oct;84(5):589-593. doi: 10.1016/j.jbspin.2016.12.008. Epub 2016 Dec 28. PMID 28039062